CLINICAL TRIAL: NCT04085224
Title: A Randomized, Open Label, Single Subcutaneous Dose 6x3 Crossover Study to Investigate the Relative Bioavailability, Safety and Tolerability Among Different Eutropin Formulations in Healthy Volunteers
Brief Title: 6x3 Crossover, Bioavailability, Safety and Tolerability Among Different Eutropin Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: LG-HGCL010
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Bioavailability, Safety and Tolerability Among Different Eutropin Formulations in Healthy Volunteers
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Somatropin
- 2 (Experimental)
  Interventions: Drug: Somatropin
- 3 (Experimental)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — LG Somatropin

SUMMARY:
A Randomized, Open Label, Single Subcutaneous Dose 6x3 Crossover Study to Investigate the Relative Bioavailability, Safety and Tolerability among Different Eutropin Formulations in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 19 or more and less than 40 years (19 =< age < 40) on the day of screening
* Negative findings in serum / urine hCG test or Subjects who are not pregnant or lactating in women

Exclusion Criteria:

* Administered other drug(s) in other clinical study within 180 days prior to the day of screening

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 2years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No